CLINICAL TRIAL: NCT02558842
Title: Intervention in the Management of Post-high Tuberculosis Hospital Through Educational Strategy and Oversight Distance in a Region With High Prevalence of the Disease: Randomized Clinical Trial
Brief Title: Intervention in the Management of Post-high Tuberculosis Hospital Through Educational Strategy and Oversight Distance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Alice Manica Muller, Principal Investigator, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 13-0192
Record Dates: First submitted 2015-09-22; First posted 2015-09-24 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Pulmonary Tuberculosis; Extra Pulmonary Tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis, Extrapulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Education Strategy (Experimental): Educational Strategy and Oversight Distance
  Interventions: Other: Education Strategy
- Routine (No Intervention): Routine hospital assistance

INTERVENTIONS:
Other: Education Strategy — Interview with the patient and their contacts, even during hospitalization, Delivering educational material about TB distribution free; Advise the patient about the BHU nearest their home, where it will follow the treatment of tuberculosis. Provide the address and telephone contact BHU this writing.
  During the time of TB treatment, contact the patient to see if it is adhering to treatment and answer questions about the disease and treatment, The contact will be performed weekly for the first month, biweekly for the other months.
  During the treatment period, contact BHU to monitor the progress of the case. Monitoring will be terminated: when the patient is discharged after cure of BHU or when the patient is absent for more than 30 days from the last scheduled visit.
  Arms: Education Strategy

SUMMARY:
Brazil ranks 17th among the 22 countries responsible for 80% of tuberculosis (TB) cases in the world. In 2010, the number of new cases of tuberculosis in Brazil was 71,930 and in 4972 RS. In 2010, Brazil had a disease incidence of 37.6 / 100,000 in 2011 fell to 36.0 / 100,000. The Rio Grande do Sul(RS)S showed an incidence rate of 46.1 / 100,000 in 2011. The mortality rate was 2.4 / 100,000 population per year in Brazil and RS.

In Porto Alegre, the incidence rate of all clinical forms of tuberculosis has remained, in the last six years, around 100/100.000 inhabitants per year, while the coefficient of pulmonary tuberculosis remained on average 50/100.000 inhabitants to year. Thus, Porto Alegre holds the 2nd place in Brazil among the capitals with the highest incidence of TB, classifying the city as high risk 5th. Porto Alegre also has a co-infection TB / HIV from 35.3% one of the highest in the country.

The best strategy to prevent new cases of tuberculosis is to invest in early diagnosis and effective treatment of existing cases of the disease. As the treatment of the disease requires daily use of medications for an extended period of time (at least 6 months), adherence becomes the main determinant of the rate of healing of disease.

There are several factors that contribute to poor adherence and treatment dropout: alcoholism, illicit drug use, infection with human immunodeficiency virus (HIV Human Immunodeficiency Virus), low education, unemployment, poor housing and prolonged the treatment. The irregular treatment and neglect are the major obstacles to the control and elimination of this disease.

Study in Porto Alegre pointed alcoholism, TB / HIV, the fact that the patient does not reside with family and low education as predictors of dropout. The dropout rate in the general population of patients with active tuberculosis was 10.7% (8.0% - 17.0%). Abandonment occurred more often within the first three meses8.

In Porto Alegre, 32.5% of new TB cases are diagnosed in hospitals. Twenty percent of these patients do not bind, after discharge, the Tuberculosis Control Program (TCP), ie, the patient egress from the hospital does not reach the basic health unit (BHU) reference for further monitoring and treatment, which is considered a serious flaw in the process control of the disease.

DETAILED DESCRIPTION:
Primary objective Test the impact on the tuberculosis cure rate of an intervention based on education and supervision from a distance in the post-discharge management of new cases diagnosed in hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be aged over 18 years.
* Diagnosis in hospital

Exclusion Criteria:

* cases where there is change in diagnosis after onset of treatment
* cases reintroduction of treatment after default
* relapse cases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2013-03; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
cure rate | proposed time of treatment (up to 24 weeks, according to the shape of the disease and the treatment used), and which has favorable performance clinical and / or radiological and / or bacteriological until the end of treatment

SECONDARY OUTCOMES:
dropout rate | it is considered abandonment cases that were without medication for more than 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Alice M Muller, MD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Alice Mânica Müller, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes